CLINICAL TRIAL: NCT02084082
Title: Bioequivalence of a Fixed Dose Combination Tablet of Linagliptin/Metformin Extended Release (5 mg/1000 mg) Compared With the Free Combination of Linagliptin and Metformin Extended Release Tablets in Healthy Subjects (an Open-label, Randomised, Single Dose, Two-way Crossover Trial)
Brief Title: Bioequivalence of a FDC Tablet of Linagliptin/Metformin (5mg/1000mg) Extended Release in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1288.9; 2013-005142-11 (EudraCT Number: EudraCT)
Record Dates: First submitted 2014-03-07; First posted 2014-03-11 (Estimated); Results first posted 2016-08-04 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2015-08

CONDITIONS: Healthy
MeSH Terms: interventions — Linagliptin; Metformin

ARMS (4):
- FDC first, fasted (Experimental): Linagliptin/Metformin ER FDC followed by single tablets of linagliptin and metformin ER, fasted condition
  Interventions: Drug: Linagliptin/Metformin ER FDC; Drug: Linagliptin; Drug: Metformin ER
- Single tablets first, fasted (Experimental): single tablets of linagliptin and metformin ER followed by Linagliptin/Metformin ER FDC, fasted condition
  Interventions: Drug: Linagliptin/Metformin ER FDC; Drug: Linagliptin; Drug: Metformin ER
- FDC first, fed (Experimental): Linagliptin/Metformin ER FDC followed by single tablets of linagliptin and metformin ER, fed condition
  Interventions: Drug: Linagliptin/Metformin ER FDC; Drug: Linagliptin; Drug: Metformin ER
- Single tablets first, fed (Experimental): single tablets of linagliptin and metformin ER followed by Linagliptin/Metformin ER FDC, fed condition
  Interventions: Drug: Linagliptin/Metformin ER FDC; Drug: Linagliptin; Drug: Metformin ER

INTERVENTIONS:
Drug: Linagliptin/Metformin ER FDC — 1x Linagliptin/Metformin FDC tablet
Drug: Linagliptin — 1x Linagliptin tablet
Drug: Metformin ER — 2x Metformin ER tablets

SUMMARY:
The purpose of this trial is to demonstrate bioequivalence of a newly developed fixed dose combination (FDC) tablet containing linagliptin and metformin extended release compared to the free combination of linagliptin and metformin extended release, both under fed and fasted conditions.

ELIGIBILITY:
Inclusion criteria:

- Healthy male or female subjects

Exclusion criteria:

- Any relevant deviation from healthy condition

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2014-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1288.9.1 Boehringer Ingelheim Investigational Site, Biberach, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study is conducted in two parts:
  Part 1 of the study was conducted in fasting conditions. Part 2 of the study was conducted in fed conditions.
Groups:
- FDC 1000 Fast/ L+M 1000 Fast: Linagliptin/Metformin Extended Release (XR) Fixed dose combination (given as 1 FDC tablet) followed by single tablets of linagliptin and metformin XR (given as 1 tablet 5 mg linagliptin and 2 tablets 500 mg metformin XR), oral with 240 mL of water after an overnight fast of at least 10 h.
  Where, L+M = Linagliptin 5mg+Metformin 1000mg
- L+M1000 Fast/ FDC1000 Fast: Single tablets of linagliptin and metformin Extended Release (given as 1 tablet 5 mg linagliptin and 2 tablets 500 mg metformin XR) followed by Linagliptin/Metformin XR Fixed Dose Combination (given as 1 FDC tablet), oral with 240 mL of water after an overnight fast of at least 10 h.
  Where, L+M = Linagliptin 5mg+Metformin 1000mg
- FDC1000 Fed/L+M1000 Fed: Linagliptin/Metformin XR FDC (given as 1 FDC tablet) followed by single tablets of linagliptin and metformin XR (given as 1 tablet 5 mg linagliptin and 2 tablets 500 mg metformin XR), oral with 240 mL of water after a high-fat, high-calorie meal.
  Where, L+M = Linagliptin 5mg+Metformin 1000mg
- L+M1000 Fed/ FDC1000 Fed: Single tablets of linagliptin and metformin XR (given as 1 tablet 5 mg linagliptin and 2 tablets 500 mg metformin XR) followed by Linagliptin/Metformin XR FDC (given as 1 FDC tablet), oral with 240 mL of water after a high-fat, high-calorie meal.
  Where, L+M = Linagliptin 5mg+Metformin 1000mg
Period: Treatment Period 1 (4 Days)
Arm/Group | FDC 1000 Fast/ L+M 1000 Fast | L+M1000 Fast/ FDC1000 Fast | FDC1000 Fed/L+M1000 Fed | L+M1000 Fed/ FDC1000 Fed
Started | 26 | 26 | 8 | 8
Completed | 26 | 26 | 8 | 8
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period 1 (35 Days)
Arm/Group | FDC 1000 Fast/ L+M 1000 Fast | L+M1000 Fast/ FDC1000 Fast | FDC1000 Fed/L+M1000 Fed | L+M1000 Fed/ FDC1000 Fed
Started | 26 | 26 | 8 | 8
Completed | 26 | 26 | 7 | 6
Not Completed | 0 | 0 | 1 | 2
Not completed — Adverse Event | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Period: Treatment Period 2 (4 Days)
Arm/Group | FDC 1000 Fast/ L+M 1000 Fast | L+M1000 Fast/ FDC1000 Fast | FDC1000 Fed/L+M1000 Fed | L+M1000 Fed/ FDC1000 Fed
Started | 26 | 26 | 7 | 6
Completed | 26 | 26 | 7 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set: All randomised subjects who received 1 dose of trial medication were included in the treated set.
Groups:
- FDC 1000 Fast or L+M 1000 Fast: The subjects in Part 1 were randomly allocated to 1 of the 2 treatment sequences T fasted_R fasted or R fasted_T fasted.
  FDC 1000 fast (T fasted): 5 mg linagliptin/1000 mg metformin XR (given as 1 FDC tablet) orally with 240 mL of water after an overnight fast of at least 10 h.
  L+M 1000 fast (R fasted): 5 mg linagliptin and 1000 mg metformin XR (given as 1 tablet 5 mg linagliptin and 2 tablets 500 mg metformin XR) oral with 240 mL of water after an overnight fast of at least 10 h.
  Where, L+M = Linagliptin 5mg+Metformin 1000mg
- FDC 1000 Fed or L+M 1000 Fed: The subjects in Part 2 were randomly allocated to 1 of the 2 treatment sequences T fed_R fed or R fed_T fed.
  FDC 1000 fed (T fed): 5 mg linagliptin/1000 mg metformin XR (given as 1 FDC tablet) orally with 240 mL of water after after a high-fat, high-calorie meal.
  L+M 1000 fed (R fed): 5 mg linagliptin and 1000 mg metformin XR (given as 1 tablet 5 mg linagliptin and 2 tablets 500 mg metformin XR) oral with 240 mL of water after a high-fat, high-calorie meal.
  Where, L+M = Linagliptin 5mg+Metformin 1000mg
- Total: Total of all reporting groups
Arm/Group | FDC 1000 Fast or L+M 1000 Fast | FDC 1000 Fed or L+M 1000 Fed | Total
Number analyzed (Participants) | 52 | 16 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.7 (10.4) | 36.1 (11.9) | 35.0 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 10 | 39
  Male | 23 | 6 | 29

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of Linagliptin in Plasma Over the Time Interval From 0 to 72 Hours (AUC0-72)
Description: AUC 0-72 (area under concentration-time curve of the Linagliptin in plasma from 0 to 72 hours) The values for geometric mean and geometric coefficient of variation (gCV) are actually adjusted geometric means and adjusted intra-individual gCVs, respectively.
Time Frame: 1 hour (h) before drug administration and 20 minutes (min), 40min, 1h,1h 30min, 2h, 3h, 4h, 5h, 6h, 8h, 10h, 12h, 24h,34h, 48h and 72h after drug administration
Population: PKS 1000 fast and PKS 1000 fed, included all treated subjects in Part 1 and Part 2, respectively, who provided at least 1 observation for at least 1 primary endpoint, without important protocol violations regarding the statistical evaluation of pharmacokinetic endpoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Groups:
- L+M 1000 Fasted: 5 mg linagliptin and 1000 mg metformin XR (given as 1 tablet 5 mg linagliptin and 2 tablets 500 mg metformin XR) oral with 240 mL of water after an overnight fast of at least 10 h.
- FDC 1000 Fasted: 5 mg linagliptin/1000 mg metformin XR (given as 1 FDC tablet) orally with 240 mL of water after an overnight fast of at least 10 h.
- L+M 1000 Fed: 5 mg linagliptin and 1000 mg metformin XR (given as 1 tablet 5 mg linagliptin and 2 tablets 500 mg metformin XR) oral with 240 mL of water after a high-fat, high-calorie meal.
- FDC 1000 Fed: 5 mg linagliptin/1000 mg metformin XR (given as 1 FDC tablet) orally with 240 mL of water after after a high-fat, high-calorie meal.
Arm/Group | L+M 1000 Fasted | FDC 1000 Fasted | L+M 1000 Fed | FDC 1000 Fed
Number analyzed (Participants) | 52 | 52 | 15 | 14
nmol*h/L | 286.639 (11.8) | 287.696 (11.8) | 234.052 (9.2) | 221.644 (9.2)
Statistical Analysis 1: Comparison: L+M 1000 Fasted vs FDC 1000 Fasted; Test type: Non-Inferiority or Equivalence — The assessment of bioequivalence was based upon 2-sided 90% confidence intervals (CIs) for the ratios of the geometric means (FDC/free combination) using an acceptance range of 80.00 to 125.00%; p < 0.0001, ANOVA; ANOVA on the logarithmic scale including effects for 'sequence', 'subjects within sequences', 'period', and 'treatment'; Adjusted Geometric Means ratio = 100.37, 90% CI 2-sided [96.562 to 104.326], Standard Error of Mean 1.023 — Ratio of (FDC 1000_fasted/ L+M 1000 fasted)
Statistical Analysis 2: Comparison: L+M 1000 Fed vs FDC 1000 Fed; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0004, ANOVA; ANOVA on the logarithmic scale including effects for 'sequence', 'subjects within sequences', 'period', and 'treatment'; Geometric mean ratio (net) = 94.70, 90% CI 2-sided [88.712 to 101.089], Standard Error of Mean 1.037 — Ratio of (FDC 1000 Fed/ L+M 1000 Fed)

2. Primary Outcome: Maximum Measured Concentration of Linagliptin in Plasma (Cmax)
Description: Cmax (maximum measured concentration of Linagliptin in plasma) The values for geometric mean and geometric coefficient of variation (gCV) are actually adjusted geometric means and adjusted intra-individual gCVs, respectively.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | L+M 1000 Fasted | FDC 1000 Fasted | L+M 1000 Fed | FDC 1000 Fed
Number analyzed (Participants) | 52 | 52 | 15 | 14
nmol/L | 8.826 (27.1) | 9.540 (27.1) | 5.791 (6.1) | 5.689 (6.1)
Statistical Analysis 1: Comparison: L+M 1000 Fasted vs FDC 1000 Fasted; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0038, ANOVA; ANOVA on the logarithmic scale including effects for 'sequence', 'subjects within sequences', 'period', and 'treatment'; Adjusted Geometric Mean ratio = 108.09, 90% CI 2-sided [99.022 to 117.989], Standard Error of Mean 1.054 — Ratio of (FDC 1000_fasted/ L+M 1000 fasted)
Statistical Analysis 2: Comparison: L+M 1000 Fed vs FDC 1000 Fed; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.0001, ANOVA; ANOVA on the logarithmic scale including effects for 'sequence', 'subjects within sequences', 'period', and 'treatment'; Adjusted Geometric Means ratio = 98.24, 90% CI 2-sided [94.067 to 102.597], Standard Error of Mean 1.024 — Ratio of (FDC 1000_fed / L+M 1000 fed)

3. Primary Outcome: Area Under the Concentration-time Curve of Metformin in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: AUC 0-t (Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point) The values for geometric mean and geometric coefficient of variation (gCV) are actually adjusted geometric means and adjusted intra-individual gCVs, respectively.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng∙h/mL
Arm/Group | L+M 1000 Fasted | FDC 1000 Fasted | L+M 1000 Fed | FDC 1000 Fed
Number analyzed (Participants) | 52 | 52 | 15 | 14
ng∙h/mL | 7146.61 (22.2) | 7146.00 (22.2) | 11326.12 (7.1) | 10980.17 (7.1)
Statistical Analysis 1: Comparison: L+M 1000 Fasted vs FDC 1000 Fasted; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.0001, ANOVA; ANOVA on the logarithmic scale including effects for 'sequence', 'subjects within sequences', 'period', and 'treatment'; Adjusted Geometric Mean ratio = 99.99, 90% CI 2-sided [93.03 to 107.47], Standard Error of Mean 1.04 — Ratio of (FDC 1000_fasted/ L+M 1000 fasted)
Statistical Analysis 2: Comparison: L+M 1000 Fed vs FDC 1000 Fed; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.0001, ANOVA; ANOVA on the logarithmic scale including effects for 'sequence', 'subjects within sequences', 'period', and 'treatment'; Adjusted Geometric Means ratio = 96.95, 90% CI 2-sided [92.24 to 101.89], Standard Error of Mean 1.03 — Ratio of (FDC 1000_fed / L+M 1000 fed)

4. Primary Outcome: Cmax of Metformin in Plasma
Description: Cmax (maximum measured concentration of the Metformin in plasma) The values for geometric mean and geometric coefficient of variation (gCV) are actually adjusted geometric means and adjusted intra-individual gCVs, respectively.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | L+M 1000 Fasted | FDC 1000 Fasted | L+M 1000 Fed | FDC 1000 Fed
Number analyzed (Participants) | 52 | 52 | 15 | 14
ng/mL | 925.709 (23.4) | 923.543 (23.4) | 947.445 (5.9) | 937.685 (5.9)
Statistical Analysis 1: Comparison: L+M 1000 Fasted vs FDC 1000 Fasted; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.0001, ANOVA; ANOVA on the logarithmic scale including effects for 'sequence', 'subjects within sequences', 'period', and 'treatment'; Adjusted Geometric Means ratio = 99.77, 90% CI 2-sided [92.464 to 107.645], Standard Error of Mean 1.046 — Ratio of (FDC 1000_fasted/ L+M 1000 fasted)
Statistical Analysis 2: Comparison: L+M 1000 Fed vs FDC 1000 Fed; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.0001, ANOVA; ANOVA on the logarithmic scale including effects for 'sequence', 'subjects within sequences', 'period', and 'treatment'; Adjusted Geometric Means ratio = 98.97, 90% CI 2-sided [94.950 to 103.160], Standard Error of Mean 1.023 — Ratio of (FDC 1000_fed / L+M 1000 fed)

5. Secondary Outcome: Area Under the Concentration-time Curve of Linagliptin in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-inf)
Description: AUC0-inf (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) for Linagliptin.
  The values for geometric mean and geometric coefficient of variation (gCV) are actually adjusted geometric means and adjusted intra-individual gCVs, respectively.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | L+M 1000 Fasted | FDC 1000 Fasted | L+M 1000 Fed | FDC 1000 Fed
Number analyzed (Participants) | 52 | 52 | 15 | 14
nmol*h/L | 461.306 (14.3) | 460.009 (14.3) | 397.945 (32.4) | 387.424 (32.4)
Statistical Analysis 1: Comparison: L+M 1000 Fasted vs FDC 1000 Fasted; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.0001, ANOVA; ANOVA on the logarithmic scale including effects for 'sequence', 'subjects within sequences', 'period', and 'treatment'; Adjusted Geometric Means ratio = 99.72, 90% CI 2-sided [95.163 to 104.493], Standard Error of Mean 1.028 — Ratio of (FDC 1000_fasted/ L+M 1000 fasted)
Statistical Analysis 2: Comparison: L+M 1000 Fed vs FDC 1000 Fed; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0778, ANOVA; ANOVA on the logarithmic scale including effects for 'sequence', 'subjects within sequences', 'period', and 'treatment'; Adjusted Geometric Means ratio = 97.36, 90% CI 2-sided [77.082 to 122.963], Standard Error of Mean 1.132 — Ratio of (FDC 1000_fed / L+M 1000 fed)

6. Secondary Outcome: AUC0-inf of Metformin in Plasma
Description: AUC0-inf(area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) for Metformin.
  The values for geometric mean and geometric coefficient of variation (gCV) are actually adjusted geometric means and adjusted intra-individual gCVs, respectively.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng∙h/mL
Arm/Group | L+M 1000 Fasted | FDC 1000 Fasted | L+M 1000 Fed | FDC 1000 Fed
Number analyzed (Participants) | 52 | 52 | 15 | 13
ng∙h/mL | 7607.75 (21.7) | 7540.21 (21.7) | 15047.37 (7.2) | 14773.59 (7.2)
Statistical Analysis 1: Comparison: L+M 1000 Fasted vs FDC 1000 Fasted; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.0001, ANOVA; ANOVA on the logarithmic scale including effects for 'sequence', 'subjects within sequences', 'period', and 'treatment'; Adjusted Geometric Means ratio = 99.11, 90% CI 2-sided [92.37 to 106.35], Standard Error of Mean 1.04 — Ratio of (FDC 1000_fasted/ L+M 1000 fasted)
Statistical Analysis 2: Comparison: L+M 1000 Fed vs FDC 1000 Fed; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.0001, ANOVA; ANOVA on the logarithmic scale including effects for 'sequence', 'subjects within sequences', 'period', and 'treatment'; Adjusted Geometric Means ratio = 98.18, 90% CI 2-sided [93.34 to 103.27], Standard Error of Mean 1.03 — Ratio of (FDC 1000_fed / L+M 1000 fed)

ADVERSE EVENTS:
Time Frame: From the first drug administration for at least 7 days after the last drug administration, up to 49 days.
Arm/Group | L+M 1000 Fasted | FDC 1000 Fasted | L+M 1000 Fed | FDC 1000 Fed
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/52 | 2/15 | 0/14
Other Adverse Events (participants affected / at risk) | 4/52 | 9/52 | 4/15 | 4/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | L+M 1000 Fasted (N=52) | FDC 1000 Fasted (N=52) | L+M 1000 Fed (N=15) | FDC 1000 Fed (N=14)
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Bone contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Muscle contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | L+M 1000 Fasted (N=52) | FDC 1000 Fasted (N=52) | L+M 1000 Fed (N=15) | FDC 1000 Fed (N=14)
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 4 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 2 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 2 | 1 | 0
Headache (Nervous system disorders) | 3 | 5 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes